CLINICAL TRIAL: NCT00331136
Title: An Open-label, Phase II, Dose-Escalation Clinical Study to Assess the Pharmacokinetics, Safety, Tolerability and Pharmacodynamics of Fixed Dose Combination of Pyronaridine and Artesunate (3:1) in Children With Acute Falciparum Malaria
Brief Title: Pyronaridine and Artesunate (3:1) in Children With Acute Uncomplicated Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry); Institute of Tropical Medicine, University of Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-003-05; NCT00329875 (obsolete NCT alias)
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: malaria; P. falciparum; artemisinin based combination therapy (ACT); antimalarial; pyronaridine artesunate (Pyramax)
MeSH Terms: conditions — Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination

ARMS (4):
- Group A (Tablets) (Experimental): Pyronaridine artesunate 6:2 mg/kg. The tablet strength is 48:16 mg oral PA, with the number of tablets depending on body weight.
  Interventions: Drug: Pyronaridine-Artesunate
- Group B (Tablets) (Experimental): Pyronaridine artesunate 9:3 mg/kg. The tablet strength is 72:24 mg oral PA, with the number of tablets depending on body weight.
  Interventions: Drug: Pyronaridine-Artesunate
- Group C (Tablets) (Experimental): Pyronaridine artesunate 12:4 mg/kg. The tablet strength is 96:32 mg oral PA, with the number of tablets depending on body weight.
  Interventions: Drug: Pyronaridine-Artesunate
- Group D (Granules) (Experimental): Pyronaridine artesunate 9:3 mg/kg. The sachet of granules strength is 60:20 mg PA, with the number of sachets depending on body weight, and is administered as a suspension with water.
  Interventions: Drug: Pyronaridine-Artesunate

INTERVENTIONS:
Drug: Pyronaridine-Artesunate — Once a day for 3 days
  Other Names: Pyramax

SUMMARY:
The purpose of this study is to evaluate three dose levels of a combination tablet and a fixed dose granule formulation of pyronaridine and artesunate (PA) for the treatment of acute uncomplicated falciparum malaria in children.

DETAILED DESCRIPTION:
This is a Phase II, open-label, sequential-group, dose-escalation, single-centre study to study pharmacokinetics, bioavailability comparison of tablets vs. granules, and safety/tolerability of PA in paediatric patients with acute symptomatic uncomplicated P. falciparum malaria. The study population will include 60 patients, comprising male and female children recruited from a single study site located in the endemic region of Gabon.

Patients will be assigned sequentially to 1 of 4 treatment groups (15 per group): Group A (Tablets) PA (48 mg + 16 mg), Group B (Tablets) PA (72 mg + 24 mg), Group C (Tablets) PA (96 mg + 32 mg), Group D (Granules) PA (60 mg + 20 mg). Oral tablets will be taken once daily for 3 consecutive days (Days 0, 1 and 2). The dose given to each patient depends on the dosing cohort group and the patient's body weight.

Each patient will attend the study site for screening and baseline procedures, as well as receipt of the first dose of study drug on Day 0 (Visit 1, baseline). Patients will be hospitalised for the first 72 hours and remain near the study site for the entire duration of the study. The patients will return to the study site for all scheduled follow-up visits until discharge on Day 42.

The primary efficacy end point for the study is the incidence of patients with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 28. In the case of adverse events reported and unresolved at Day 42, patients will be followed up for a further 30 days, or until resolution of the event.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with symptoms of acute uncomplicated falciparum malaria with the following inclusion criteria:

* Male or female children, being between 2 and 14 years of age inclusive
* Weight between 10 and 40 kg inclusive
* Written informed consent, in accordance to local practice, provided by parent/guardian. If the parent/guardian is unable to write, witnessed consent is permitted according to local ethical considerations. Where possible, parent assent will be sought
* Absence of severe malnutrition (defined as mid upper arm circumference <110mm)
* Presence of acute symptomatic uncomplicated P. falciparum malaria with a diagnosis confirmed by a positive blood smear with asexual forms of P. falciparum only (i.e. no mixed infection) plus measured temperature of ≥37.5°C (depending on method of measurement as below) or history of fever within the past 24 hours :
* the acceptable range is between 1,000 and 200,000 asexual parasite count/μl of blood and
* axillary/tympanic temperature of ≥37.5°C or oral/rectal temperature of ≥38.0°C
* Females of childbearing potential are not allowed to be pregnant or lactating and must be willing to use adequate measures of contraception during the study period
* Ability to comply with the study visit schedule and the study protocol for the duration of the study

Exclusion Criteria:

* Patients with signs and symptoms of severe/complicated malaria requiring parenteral antimalarial treatment according to the WHO Criteria 2000
* Mixed Plasmodium infection
* Severe vomiting, defined as >3 times in the 24 hours prior to inclusion in the study or inability to tolerate oral treatment, or severe diarrhoea defined as >3 watery stools per day
* Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, acute QTc interval greater or equal to 450 msec), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other abnormality (including head trauma)
* Presence of febrile conditions caused by diseases other than malaria
* Known history of hypersensitivity, allergic or adverse reactions to pyronaridine or artesunate or other artemisinins
* Use of any other antimalarial treatment within 2 weeks prior to start of the study as confirmed by Lignin test and Saker Solomon urine test
* For females of childbearing potential, positive urine pregnancy test or lactating
* Use of an investigational drug within the past 8 weeks
* Known active Hep A immunoglobulin, Hep B surface antigen, or Hep C antibody
* Known seropositive HIV antibody
* Liver function tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] levels) >3 times the upper limit of normal
* Known significant renal impairment as indicated by a serum creatinine ≥2 mg/dL
* Previous participation in this clinical study

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ramharter, MD, Principal Investigator — Albert Schweitzer Hospital, Lambaréné, Gabon
Locations (1):
- Medical Research Unit, Albert Schweitzer Hospital, Lambaréné, Gabon

REFERENCES:
- [Background] Ringwald P, Bickii J, Basco L. Randomised trial of pyronaridine versus chloroquine for acute uncomplicated falciparum malaria in Africa. Lancet. 1996 Jan 6;347(8993):24-8. doi: 10.1016/s0140-6736(96)91558-5. PMID 8531545
- [Derived] Ramharter M, Djimde AA, Borghini-Fuhrer I, Miller R, Shin J, Aspinall A, Richardson N, Wibberg M, Fleckenstein L, Arbe-Barnes S, Duparc S. Safety and efficacy of pyronaridine-artesunate paediatric granules in the treatment of uncomplicated malaria in children: insights from randomized clinical trials and a real-world study. Malar J. 2024 Feb 28;23(1):61. doi: 10.1186/s12936-024-04885-3. PMID 38418982
- [Derived] Ayyoub A, Methaneethorn J, Ramharter M, Djimde AA, Tekete M, Duparc S, Borghini-Fuhrer I, Shin JS, Fleckenstein L. Population Pharmacokinetics of Pyronaridine in Pediatric Malaria Patients. Antimicrob Agents Chemother. 2015 Dec 14;60(3):1450-8. doi: 10.1128/AAC.02004-15. PMID 26666916
- [Derived] Duparc S, Borghini-Fuhrer I, Craft CJ, Arbe-Barnes S, Miller RM, Shin CS, Fleckenstein L. Safety and efficacy of pyronaridine-artesunate in uncomplicated acute malaria: an integrated analysis of individual patient data from six randomized clinical trials. Malar J. 2013 Feb 21;12:70. doi: 10.1186/1475-2875-12-70. PMID 23433102
- [Derived] Ramharter M, Kurth F, Schreier AC, Nemeth J, Glasenapp Iv, Belard S, Schlie M, Kammer J, Koumba PK, Cisse B, Mordmuller B, Lell B, Issifou S, Oeuvray C, Fleckenstein L, Kremsner PG. Fixed-dose pyronaridine-artesunate combination for treatment of uncomplicated falciparum malaria in pediatric patients in Gabon. J Infect Dis. 2008 Sep 15;198(6):911-9. doi: 10.1086/591096. PMID 18694333
- See also: Shin Poong Pharmaceuticals — http://www.shinpoong.co.kr/

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Tablets): Pyronaridine artesunate 6:2 mg/kg. Number of PA tablets (48 mg + 16 mg) administered based on posology. 3-day course of once-daily dosing.
- Group B (Tablets): Pyronaridine artesunate 9:3 mg/kg. Number of PA tablets (72 mg + 24 mg) administered based on posology. 3-day course of once-daily dosing.
- Group C (Tablets): Pyronaridine artesunate 12:4 mg/kg. Number of PA tablets (96 mg + 32 mg) administered based on posology. 3-day course of once-daily dosing.
- Group D (Granules): Pyronaridine artesunate 9:3 mg/kg. Number of PA sachets containing granules (60 mg + 20 mg) administered based on posology. Sachet is administered as a suspension with water. 3-day course of once-daily dosing.
Period: Overall Study
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Started | 15 | 15 | 15 | 15
Completed | 10 | 8 | 15 | 14
Not Completed | 5 | 7 | 0 | 1
Not completed — Adverse Event | 3 | 5 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Not treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all subjects who received at least 1 dose of study drug. Males/Females between ages of 2 and 14 years, with body weight between 10 and 40kg.
Groups:
- Group A (Tablets): Pyronaridine artesunate 6:2 mg/kg
- Group B (Tablets); Group D (Granules): Pyronaridine artesunate 9:3 mg/kg
- Group C (Tablets): Pyronaridine artesunate 12:4 mg/kg
- Total: Total of all reporting groups
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules) | Total
Number analyzed (Participants) | 14 | 15 | 15 | 15 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (2.19) | 5.9 (3.48) | 5.8 (2.60) | 4.6 (1.96) | 5.5 (2.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 9 | 7 | 29
  Male | 8 | 8 | 6 | 8 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 14 | 15 | 15 | 15 | 59
Height [Mean (Standard Deviation); unit: cm] | 110.4 (13.16) | 109.3 (18.66) | 111.8 (16.08) | 103.3 (14.31) | 108.7 (15.67)
Weight [Mean (Standard Deviation); unit: kg] | 18.7 (5.54) | 18.8 (7.00) | 19.0 (6.44) | 16.5 (5.15) | 18.2 (6.01)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With PCR-corrected Adequate Clinical and Parasitological Response (ACPR) on Day 28
Description: Clearance of asexual parasitaemia within 7 days of initiation of study medication without recrudescence within 28 days, without previously meeting any of the criteria for early treatment failure, late clinical failure, or late parasitological failure.
Time Frame: Day 28
Population: Per protocol population: all patients who received a full course of study treatment, had a known status of the primary efficacy variable, and did not have major protocol violations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 11 | 13 | 15 | 14
Participants | 11 | 13 | 15 | 14

2. Secondary Outcome: Parasite Clearance Time
Description: The time from first dosing to the time of first blood draw with parasite clearance. Parasite clearance is defined as zero presence of parasites for 2 consecutive negative readings taken between 8 and 24 hours apart.
Time Frame: Day 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 11 | 13 | 15 | 14
hours | 16.4 [16.1 to 22.4] | 16.1 [8.3 to 16.4] | 8.1 [8.0 to 16.0] | 8.3 [8.1 to 15.9]

3. Secondary Outcome: Treatment Success or Failure
Description: Treatment success for the ACPR analysis is defined as the clearance of asexual parasitaemia within 7 days of initiation of study medication without recrudescence within 28 days, without previously meeting any of the criteria for early treatment failure, late clinical failure, or late parasitological failure. Early and late failures are classified according to the WHO Protocol 2005.
Time Frame: Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 11 | 13 | 15 | 14
Participants
  Treatment success | 11 | 13 | 15 | 14
  Treatment failure | 0 | 0 | 0 | 0

4. Secondary Outcome: Fever Clearance Time
Description: The time from first dosing to the first normal reading with fever clearance, defined as 2 consecutive assessments without fever (<37.5°C) taken between 8 and 24 hours apart.
  NB: Time to fever clearance was only summarised for subjects who had fever at baseline or within the first 24 hours after the start of study treatment. Since only 12 subjects in total had fever during this time, the time to fever clearance estimates are not very meaningful.
Time Frame: Day 3
Population: Only patients with a fever at baseline or within 24 hours were taken into account.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 3 | 5 | 3 | 1
hours | 8.2 [8.1 to 16.2] | 8.6 [8.1 to 17.2] | 8.2 [8.1 to 16.2] | 8.2 [NA to NA] — Data available for only one participant, therefore, it is not possible to calculate the 95% Confidence Interval

5. Secondary Outcome: Number of Patients With PCR-corrected ACPR on Day 14
Description: Clearance of asexual parasitaemia within 7 days of initiation of study medication without recrudescence within 14 days.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 11 | 13 | 15 | 14
Participants | 11 | 13 | 15 | 14

6. Secondary Outcome: Number of Patients With Parasite Clearance at Day 1, 2 and 3
Description: Zero presence of parasites for 2 consecutive negative readings taken between 8 and 24 hours apart.
Time Frame: Days 1, 2, 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 11 | 13 | 15 | 14
Participants
  Clearance by >0 - 24 hours (Day 1) | 10 | 11 | 14 | 14
  Clearance by >24 - 48 hours (Day 2) | 1 | 2 | 1 | 0
  Clearance by >48 - 72 hours (Day 3) | 0 | 0 | 0 | 0
  Clearance by >72 hours (Day 3 onwards) | 0 | 0 | 0 | 0
  No clearance achieved | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With P. Falciparum Gametocytes During the Trial
Description: The number of gametocytes per μl at Days 0, 3, 7, 14, 21, 28, 35, and 42 summarised from blood slides taken on the respective days.
  P. falciparum gametocytes are responsible for transmission from host to vector.
Time Frame: Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 11 | 13 | 15 | 14
Participants
  Baseline | 2 | 0 | 1 | 1
  >0-24 hours | 3 | 1 | 1 | 1
  >24-48 hours | 2 | 0 | 0 | 0
  >48-72 hours | 2 | 1 | 0 | 0
  >72 hours - Day 7 | 2 | 0 | 1 | 0
  >Day 7 - Day 28 | 1 | 0 | 0 | 0
  >Day 28 - Day 42 | 0 | 0 | 0 | 0
  >Day 42 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Patients With Fever Clearance at Day 1, 2 and 3
Description: Patient without fever for 2 consecutive readings taken between 8 and 24 hours apart.
  NB: Percentage of fever clearance was only summarised for subjects who had fever at baseline or within the first 24 hours after the start of study treatment. Since only 12 subjects in total had fever during this time, the time to fever clearance estimates are not very meaningful.
Time Frame: Days 1, 2, 3
Population: Only patients with a fever at baseline or within 24 hours were taken into account.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 3 | 5 | 3 | 1
Participants
  Clearance by >0 - 24 hours | 3 | 5 | 3 | 1
  Clearance by >24 - 48 hours | 0 | 0 | 0 | 0
  Clearance by >48 - 72 hours | 0 | 0 | 0 | 0
  No clearance achieved | 0 | 0 | 0 | 0

9. Secondary Outcome: Crude ACPR on Day 14, 28 and 42
Description: The proportion of patients with crude (non-PCR corrected) ACPR.
Time Frame: Days 14, 28, 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 11 | 13 | 15 | 14
Participants
  Day 14 | 11 | 13 | 15 | 14
  Day 28 | 11 | 10 | 15 | 14
  Day 42: number analyzed (Participants) | 10 | 12 | 15 | 14
  Day 42 | 7 | 6 | 13 | 12

10. Secondary Outcome: Number of Patients With PCR-corrected ACPR on Day 42
Description: Clearance of asexual parasitaemia within 7 days of initiation of study medication without recrudescence within 42 days.
Time Frame: Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
Number analyzed (Participants) | 10 | 9 | 15 | 14
Participants | 10 | 8 | 15 | 13

ADVERSE EVENTS:
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Arm/Group | Group A (Tablets) | Group B (Tablets) | Group C (Tablets) | Group D (Granules)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 13/14 | 11/15 | 13/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Tablets) (N=14) | Group B (Tablets) (N=15) | Group C (Tablets) (N=15) | Group D (Granules) (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1.7% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Tablets) (N=14) | Group B (Tablets) (N=15) | Group C (Tablets) (N=15) | Group D (Granules) (N=15)
Plasmodium falciparum infection (Infections and infestations) | 1 | 6 | 2 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 3 | 5
Ascariasis (Infections and infestations) | 1 | 1 | 3 | 1
Malaria (Infections and infestations) | 4 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 2 | 1
Abscess (Infections and infestations) | 1 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 2
Giardiasis (Infections and infestations) | 0 | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Schistosomiasis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 1 | 2 | 1
Fatigue (General disorders) | 1 | 2 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No